CLINICAL TRIAL: NCT06743737
Title: Sensitivity and Specificity Study of Electromedical Device Nexkin DSPT and Manual Measurement of Hives in Allergy Skin Prick Tests
Brief Title: Digital Device Reading Skin Prick Test
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: sitem-insel AG Bern (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-D0059
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Allergy Skin Prick Test Reading

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Digital skin test reading device — The device to be studied measures optically the size of the wheals from skin tests (SPT) performed for the diagnosis of allergen sensitization.

SUMMARY:
Skin prick tests (SPTs), or intraepidermal tests, are the first diagnostic approach for people with a suspected allergy. SPTs are very simple, safe and quick. They are cheap tests and are very useful as a screening test for allergy, especially in diseases like bronchial asthma, rhinoconjunctivitis, food/drug allergy and anaphylaxis. Together with the clinical history, SPTs allow to draw conclusions on allergies based on the sensitization pattern.

Nevertheless, the technique itself has evolved very little and continues to be performed entirely manually. This has a few drawbacks that limit the utility of the tests, in many cases limiting them to a purely qualitative assessment.

In comparison to standard practice (manual measurement), the digital skin test reading device Nexkin DSPT can provide the following benefits for project participants: Automates and digitizes the test reading, provides test results in digital format, reduces variability and subjectivity and greater consistency of diagnosis, reduces manual tasks allowing health professionals providing quantitative instead of qualitative results and avoiding potential human errors and allows a faster workflow, resulting in shorter patient visits.

The aim of this study is to validate the clinical utility of the electromedical skin test reading device Nexkin DSPT regarding its use in allergology clinics for the reading of skin prick allergy tests. The overall purpose of the study is to determine the sensitivity and specificity of skin prick tests (SPT) performed using the current practice of the fully manual SPT procedure and those performed using the Nexkin SPT DSPT (digital) procedure and to compare the sensitivity and specificity of both methods.

ELIGIBILITY:
Inclusion Criteria:

Patients who will undergo skin prick tests with panels of aeroallergens and/or foods.

Over 18 years of age. The patient or their representative has given consent to participate in the study.

The patient must not have taken an antihistamine in the last 5 days.

Exclusion Criteria:

Patients who are evaluated by more than 40 prick tests. Patients who have taken an antihistamine within the previous 5 days. Patients who are being treated with antidepressants or other drugs with an antihistamine effect.

Patients who suffer severe atopic dermatitis with forearm involvement. Patients with dermographism. Patients who are evaluated by intradermal testing. Pregnant women or women suspected to be pregnant. Vulnerable patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with a food or aeroallergy who require a SPT in the routine allergy workup are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of the histamine (positive control) wheal by healthcare professional | At enrollment
Measurement of the NaCl (negative control) wheal by healthcare professional | At enrollment
Measurement of the histamine (positive control) wheal by digital device | At enrollment
Measurement of the NaCl (negative control) wheal by digital device | At enrollment

SECONDARY OUTCOMES:
Measure of the time involved in the complete reading and recording of the results | At enrollment
  Minutes and seconds of procedure (testing & recording of results) will be recorded for both the manual procedure and the procedure using the digital device

CONTACTS AND LOCATIONS:
Overall Officials: Elnaz Arjmand, Principal Investigator — Inselspital, Bern / sitem-Insel AG
Locations (1):
- Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR